CLINICAL TRIAL: NCT07364695
Title: Early Postoperative Function After Open Versus Ultrasound-Guided Trigger Finger Release: A Prospective Comparative Cohort Study
Brief Title: Early Postoperative Function After Open Versus Ultrasound-Guided Trigger Finger Release
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Rohit Garg, Director, Hand Surgery Fellowship Program, Assistant Professor of Orthopedic Surgery, Massachusetts General Hospital
Other Study IDs: 2023P003220
Record Dates: First submitted 2025-12-11; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Trigger Finger
Keywords: trigger finger release; ultrasound; open; clinical outcomes; return to work
MeSH Terms: conditions — Trigger Finger Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Open Release: Patients who underwent open trigger finger release
- Ultrasound-Guided Release: Patients who underwent ultrasound-guided trigger finger release
  Interventions: Device: UltraGuideTFR (Sonex Health, MN, USA)

INTERVENTIONS:
Device: UltraGuideTFR (Sonex Health, MN, USA) — SonexHealth percutaneous trigger finger release device used in ultrasound-guided release cohort
  Groups: Ultrasound-Guided Release

SUMMARY:
Clinical outcomes after open trigger finger release are excellent. Minimally invasive techiques with ultrasound guidance theoretically offer advantages for faster recovery but this technique has not been compared prospectively with the standard of care (open trigger release). This study aims to prospectively analyze patient-reported outcomes in patients undergoing open vs. ultrasound-guided trigger finger release.

DETAILED DESCRIPTION:
Trigger finger is initially treated conservatively. Conservative treatment options include modification of activities, painkiller administration, splinting, and corticosteroid injections (1). Open or minimally invasive surgical treatment can be considered if conservative treatment fails. Minimally invasive surgery options consist of ultrasound-guided or blind percutaneous trigger finger release.

Many studies have reported good clinical outcomes after ultrasound-guided trigger finger release, including low rates of catching or locking recurrence rates, high QuickDASH scores and high patient satisfaction (2-4).

Postoperative clinical outcomes of open surgery have been widely compared to percutaneous surgery (5-8). However, the comparison of postoperative results between ultrasound-guided and open trigger finger release has been scarcely reported. Nikolaou et al. reported that ultrasound-guided trigger finger release resulted in a significantly sooner return to normal activities and better patient-reported cosmetic outcomes than open trigger finger release (9). Success rates and mean QuickDASH scores did not differ significantly between these groups in this cohort.

The potential benefits of ultrasound-guided trigger finger release compared to open trigger finger release have yet to be investigated. This study aims to prospectively analyze patient-reported outcomes in patients undergoing open vs. ultrasound-guided trigger finger release.

ELIGIBILITY:
Inclusion Criteria:

* undergoing trigger finger release for the index through small fingers due to symptoms refractory to conservative treatment and elected for surgical intervention through shared decision-making
* English-speaking adults (≥18 years of age)
* Patients with inflammatory arthritis were included if their diagnosis had been established ≥5 years prior without exacerbations in the past 5 years. Those on immunomodulatory therapy were required to have been on a stable regimen for ≥5 years without flare-ups.

Exclusion Criteria:

* prior surgery on the affected finger
* corticosteroid injection in the affected hand within 6 weeks
* additional hand or wrist pathology requiring concurrent surgery
* symptomatic trigger finger in the contralateral extremity
* prior surgical pulley release in either hand within 6 months of enrollment
* Systemic inflammatory disease (e.g., rheumatoid arthritis, lupus) not controlled
* inflammatory arthritis if diagnosis established <5 years, exacerbation within the past 5 years, or modifications to immunomodulatory therapy within 5 years of enrollment
* Amyloidosis
* Diabetes not controlled by a stable dose of medication over the past three months
* Pregnant or planning pregnancy in the next 6 months
* Workers' compensation subjects
* Inability to provide a legally acceptable Informed Consent Form and/or comply with all follow-up requirements, including patients who do not speak English
* other medical, social, or psychological conditions that, in the opinion of the investigator, preclude them from receiving the pre-treatment, required treatment, and post-treatment procedures and evaluations.
* Trigger Thumb

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing trigger finger release for the index through small fingers was conducted from June 2023 through June 2024 at two tertiary care academic medical centers in an integrated health network
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2023-06-20 (Actual); Primary Completion 2024-06-26 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Activities of Daily Living (Study-specific questionnaire) | From enrollment to final follow-up at 6 months
  Study-specific survey of limitations with Activities of Daily Living. Responses for questions on the study-specific survey for limitations with ADLS utilized a Likert scale with 1 representing no difficulty with the task and 5 being unable to perform the task due to limitations from trigger finger symptoms. Likert scale responses for the 12 ADLs on the survey were summated for final scores ranging from 14 (no difficulty with any ADLs) to 70 (unable to perform any ADLs). These were standardized to a 100-point scale to facilitate clinical interpretation of outcomes. A score of 0 represented no functional limitations with ADLs and a score of 100 represented inability to perform any ADL on the survey.
Pain on the Visual Analogue Scale | From enrollment to final follow-up at 6 months
  VAS pain score on a scale from 1 to 10 with a score of 1 representating no pain and score or 10 representing maximal pain.

SECONDARY OUTCOMES:
Timing of Return to work | From 2 days post-procedure to final follow-up at 6 months
  Timing of return to work in days as reported by patient. Minimum value is 0 days, meaning patient reported returning to work on the day of the procedure. No maximum value applicable.
Patient satisfaction with procedure | Single evaluation at final follow-up 6 months post-procedure
  Patient reported satisfaction with procedure. Response of either yes or no to the following question: Are you satisfied with the procedure, and would you choose to have it again for a similar problem?

OTHER OUTCOMES:
Proximal interphalangeal joint (PIPJ) flexion | Assessments at the preoperative and two-week follow-up visits
  Proximal interphalangeal (PIP) flexion measured with a goniometer and recorded in degrees. Minimum and maximum values within physiologic range of motion for the PIPJ.
PIPJ motion as evaluated by distance from fingertip to distal palmar crease in composite flexion | Assessments at the preoperative and two-week follow-up visits
  Distance in millimeters from fingertip to the distal palmar crease (DPC) in composite flexion. Minimum of 0 cm, maximum value of >5 cm which represents absence of functionally meaningful finger flexion.
PIPJ flexion contracture (if present) | Assessments at the preoperative and two-week follow-up visits
  If present, PIPJ flexion contracture measured using a goniometer and recorded in degrees. Minimum value of 0 degrees representing absence of flexion contracture, maximum value within physiologic range of motion for the PIPJ.
Analegesia requirement | From enrollment to final follow-up at 6 months
  Pain medication requirement including acetaminophen, anti-inflammatories, and/or narcotics. Open response from patients for the following question: How many oxycodone or other narcotic medications are you taking post-op?
Grip Strength | Assessments at the preoperative and two week follow-up visits
  Grip strength was evaluated using a Jamar dynamometer setting #2.

CONTACTS AND LOCATIONS:
Overall Officials: Rohit Garg, MBBS, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
Anonymized patient data can be shared upon reasonable request for transparency
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: January 2023 through January 2027
Access Criteria: De-identified IPD will be available to qualified researchers who submit a methodologically sound proposal. Requests may be made to the principal investigator. Access will be provided through a secure data-sharing platform following execution of a data use agreement

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-06-06): https://cdn.clinicaltrials.gov/large-docs/95/NCT07364695/Prot_SAP_ICF_000.pdf